CLINICAL TRIAL: NCT04701450
Title: Questionnaire Study to Evaluate Patient Satisfaction Between Digital, Telephonic and Conventional Obtaining of Consent for Anaesthesia
Brief Title: Evaluation of Digital, Telephonic and Conventional Consent for Anaesthesia
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, David M Baron, MD, PhD, Assoc. Prof. PD Dr. David Baron, EDIC, Medical University of Vienna
Other Study IDs: 1688/2018
Record Dates: First submitted 2021-01-01; First posted 2021-01-08 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- conventional: consent for anaesthesia is obtained as part of a conversation with physical attendance
- telephonic: consent for anaesthesia is obtained telephonically
- digital: a digital survey and video information is used to inform the patient about the anaesthetic procedure
  Interventions: Other: digital consent

INTERVENTIONS:
Other: digital consent — the patient's medical history is taken in a digital survey, information about the anaesthetic procedure is aided by video material
  Groups: digital

SUMMARY:
In this study, the investigators aim to evaluate patient satisfaction between three methods of obtaining informed consent for anaesthesia. Patients are asked to partake in a short survey after being informed about the anaesthetic procedure either conventionally in the anesthesia department, telephonically or digitally.

DETAILED DESCRIPTION:
Patient satisfaction plays an important role to improve the process of medical procedures as well as patient outcome. Evaluating the subjectively experienced satisfaction is challenging. The investigators will use a questionnaire and assess waiting times in the process to determine patient satisfaction between digital, telephonic and conventional obtaining of informed consent for anaesthesia.

In this questionnaire study, patients are asked to partake in a survey after the process of obtaining consent for anaesthesia is completed. The questionnaire covers aspects of patient satisfaction with the process, such as subjective assessment of comprehensibility, waiting time and privacy.

Patients are divided into three groups. In one group, consent is obtained conventionally, in form of a visit to our anaesthesia department. In the other two groups, consent is obtained telephonically and digitally, respectively. Patients are not randomised into these groups, but included into the study after the process of obtaining consent by one of the three methods mentioned above is completed.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom consent for anaesthesia is obtained

Exclusion Criteria:

* Age < 18 years
* Language barrier
* Patients with appointed legal guardians
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients for whom consent for anaesthesia is obtained for an elective procedure
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction after informed consent | Immediately after obtaining informed consent
  Assessment of subjectively experienced satisfaction with the process of obtaining informed consent for anesthesia

SECONDARY OUTCOMES:
Overall waiting time of patients | Up to three hours; from administration for informed consent until completion of informed consent
  Patient's overall waiting time in the process of obtaining consent
Time expense of informed consent | Up to 60 minutes; from start until end of informed consent
  Overall time expense for the anaesthesiologist who is connsenting the patient
Intraoperative complications | Up to 12 hours; From start until end of the planned surgical procedure
  Incidence of unexpected medical complications during the surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: David M. Baron, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Vienna General Hospital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No